CLINICAL TRIAL: NCT00349570
Title: Xtract™ Aspiration Catheter Registry Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumen Biomedical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90-1027
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Fresh Soft Emboli or Thrombi in the Arteries.
Keywords: thrombus; aspiration catheter
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Xtract Aspiration Catheter

SUMMARY:
Intra-coronary thrombosis and thromboembolism continues to be a challenge for percutaneous coronary and other vascular interventional techniques. The Xtract™ Aspiration Catheter is a single use device designed to remove fresh, soft emboli and thrombi from the arterial system using standard catheter techniques, compatible with 6 Fr guide catheters and 0.014 guidewires. The purpose of this registry study is to validate the design and demonstrate the performance of the Xtract Aspiration Catheter as a thrombectomy catheter during percutaneous intervention of vessels in the arterial system. Subjects will be enrolled during percutaneous intervention when the Interventional Physician decides a thrombectomy catheter is needed to remove thrombus during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Planned percutaneous intervention to a native coronary, coronary vein graft, renal artery or carotid artery lesion
* Angiographic evidence of thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-08; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study will be to evaluate the performance of the Xtract Aspiration Catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Webster, MD, Principal Investigator — Auckland City Hospital
Locations (2):
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - ChristChurch Hospital, Christchurch